CLINICAL TRIAL: NCT06195345
Title: Individual Cerebral Hemodynamic Oxygenation Relationships (ICHOR 1)
Acronym: ICHOR 1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Matthew Borzage, USC Faculty/ Non Physician CWR, Children's Hospital Los Angeles
Other Study IDs: CHLA-18-00439
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: HIE; TBI (Traumatic Brain Injury); TBI; Hemodynamic Instability; Hypoxic-Ischemic Encephalopathy
MeSH Terms: conditions — Brain Injuries, Traumatic; Hypoxia-Ischemia, Brain | interventions — Magnetic Resonance Imaging; Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pediatric Patients: Children scheduled for clinical MR imaging.
  Interventions: Diagnostic Test: MR Imaging

INTERVENTIONS:
Diagnostic Test: MR Imaging — MR imaging pertaining to the patient and project (ICHOR 1)
  Other Names: MRI; Medical Imaging

SUMMARY:
This is an observational study in patients who require clinical anesthesia. The main purpose of this study is to understand whether there are differences in the cerebral blood flow, and oxygen metabolism affected by different types of anesthesia. Subjects who require clinical anesthesia for a clinical MRI and for whom the use of anesthetics for the exam are in clinical equipoise are asked to join the study. All eligible subjects will be asked to provide informed consent before participating in the study.

DETAILED DESCRIPTION:
This is an observational study in patients who require clinical anesthesia. The main purpose of this study is to understand whether there are differences in the cerebral blood flow, and oxygen metabolism affected by different types of anesthesia. Subjects who require clinical anesthesia for a clinical MRI and for whom the use of anesthetics for the exam are in clinical equipoise are asked to join the study. All eligible subjects will be asked to provide informed consent before participating in the study.

Treatment:

Those who meet eligibility criteria, and who undergo the informed consent, will have their MRI extended by up to 7.5 minutes for up to 5 times. Standard-of-care anesthesia safety, dose and monitoring will not be changed. During their MRI, the additional images acquired will teach us about cerebral blood flow and cerebral venous oxygenation. Participants will also have non-invasive monitoring of their hematocrit immediately following the exam.

Safety Assessment:

The experiment will occur in the standard-of-care clinical MRI environment. All patient safety and monitoring will remain in place. Throughout the induction, maintenance and recovery from anesthesia, all procedures will occur in the standard of care environment and will be overseen by trained clinical personnel.

Efficacy Assessment:

Structural, and/or cerebral blood flow and/or metabolism MRIs will be collected from all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are able to tolerate an MRI.
* Are patients scheduled for a clinically indicated MRI.
* Between birth and up to 18 years.

Exclusion Criteria:

* Presence of an MRI-incompatible device or implant (e.g. pacemakers, stents)
* Unable to tolerate the enclosed spaces and loud noises for the duration of time in scanner required to obtain an MRI.
* Preterm infants less than 25 weeks
* Any patient who is clinically too unstable to extend their MRI by up-to 7.5 minutes.

Ages: 1 Minute to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Neonates and young children
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change in cerebral blood flow (ml blood/100g/min) | Time points over which the change is assessed: change from (1) start of MRI, through (2) MRI completion, an average of 60 minutes.
  Phase contrast (PC) acquisition via MRI will be used to assess any impact of anesthesia on cerebral blood flow.
Change in cerebral metabolic rate of oxygen (ml O2/100g/min) | Time points over which the change is assessed: change from (1) start of MRI, through (2) MRI completion, an average of 60 minutes.
  T2 relaxation under spin tagging (TRUST) acquisition via MRI will be used to assess any impact of anesthesia on cerebral metabolic rate of oxygen.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes